CLINICAL TRIAL: NCT03605186
Title: Prevention of Oral Mucositis After Using Chamomile Oral Cryotherapy Versus Oral Cryotherapy in Pediatric Cancer Patients Receiving Chemotherapy: (A Randomized Pilot Study)
Brief Title: Prevention of Oral Mucositis After Using Chamomile Oral Cryotherapy Versus Oral Cryotherapy in Pediatric Cancer Patients Receiving Chemotherapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Dina Yousef Abdel Aleem Essa, Master Degree Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-07-08
Record Dates: First submitted 2018-07-11; First posted 2018-07-30 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Oral Mucositis (Ulcerative) Due to Antineoplastic Therapy
Keywords: chamomile cryotherapy; cryotherapy; cancer; children; pediatric; chemotherapy
MeSH Terms: conditions — Stomatitis; Ulcer; Neoplasms | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chamomile oral cryotherapy (Experimental): 1. The infusion of chamomile will be prepared in the clinic with 400 mL of distilled water and 10 g of chamomile flowers (Chamomile classic infusion, Royal Herbs).
  2. Ice cubes will be prepared in special ice trays placed in the chemotherapy center for this purpose.
  3. Patient will receive a cup of ice cubes which is continuously replenished before being emptied.
  4. Patients will be instructed to swish the ice cubes around their oral cavities starting 5 minutes before chemotherapy infusion, continuing 30 minutes throughout the session and for additional 35 minutes after completion of intravenous chemotherapy session.
  Interventions: Other: Chamomile oral cryotherapy
- Oral cryotherapy (Active Comparator): 1. The plain icecubes will be prepared in the clinic with 400 mL of distilled water.
  2. Ice cubes will be prepared in special ice trays placed in the chemotherapy center for this purpose.
  3. Patient will receive a cup of ice cubes which is continuously replenished before being emptied.
  4. Patients will be instructed to swish the ice cubes around their oral cavities starting 5 minutes before chemotherapy infusion, continuing 30 minutes throughout the session and for additional 35 minutes after completion of intravenous chemotherapy session.
  Interventions: Other: Oral cryotherapy

INTERVENTIONS:
Other: Chamomile oral cryotherapy — The infusion of chamomile will be prepared in the clinic with 400 mL of distilled water and 10 g of chamomile flowers (Chamomile classic infusion, Royal Herbs). Patients are asked to swish the chamomile ice cubes around their oral cavities starting 5 minutes before chemotherapy infusion, continuing 30 minutes throughout the session and for additional 35 minutes after completion of intravenous chemotherapy session.
  Other Names: chamomile oral infusion
  Arms: Chamomile oral cryotherapy
Other: Oral cryotherapy — The plain icecubes will be prepared in the clinic with 400 mL of distilled water. Patients are asked to swish the ice cubes around their oral cavities starting 5 minutes before chemotherapy infusion, continuing 30 minutes throughout the session and for additional 35 minutes after completion of intravenous chemotherapy session.
  Arms: Oral cryotherapy

SUMMARY:
oral mucositis is a painful situation that significantly affects patients' quality of life with the severe cases being associated with ulcerated mucosa and secondary infection which may lead to life-threatening sepsis.Chamomile infusion in cryotherapy was used to aid in reduction of chemotherapy induced mucositis and to enhance the effect of standard cryotherapy alone by its anti-inflammatory, antifungal and antibacterial effect. The occurrence of oral mucositis is a significant complication of chemotherapy with prevalence of up to 80% in pediatric patients.The study is to be conducted at the in and outpatient clinics at the Department of Pediatric Oncology, National Cancer Institute,Egypt. A Structured interview questionnaire sheet will be filled with personal, medical and dental history. Intraoral examination will be carried out using sterile latex gloves, masks, plain mouth mirrors, sterile gauze and wooden tongue depressor. Patients who will agree to participate in the study will watch a video explaining how to perform oral hygiene.Preparation of the interventions is done in the clinic with 400 ml of distilled water with or without the infusion of 10 g of chamomile flowers."Chamomile classic infusion, Royal Herbs" .Ice cubes will be prepared in special ice trays placed in the chemotherapy center for this purpose.Patients will be instructed to swish the ice cubes around their oral cavities starting 5 minutes before chemotherapy infusion, continuing 30 minutes throughout the session and for additional 35 minutes after completion of intravenous chemotherapy session. Follow ups are done at the 8th,15th and the 21st day of interventions application.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy and intact oral mucosa.
2. Patients diagnosed with bone tumor (osteosarcoma) for the first time.
3. Patients receiving Methotrexate as part of their chemotherapeutic regimen.
4. Both male and female patients undergoing chemotherapy at In and Out patient units of Pediatric Oncology department.
5. Age of patient ranging (6- 18) years old.
6. Legal representatives of patient must be able to read, understand and provide informed consent to participate in the trial.
7. Patients with no history of dental discomfort related to cold or hot food or beverage intake.

Exclusion Criteria:

1. Administration of antiviral or antifungal therapy and/or any other treatment for oral mucositis before enrollment in the study.
2. Presence of advanced or severe periodontitis (pocket depth more than 6mm).
3. Patients who were supposed to receive head and neck radiotherapy as part of their treatment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in "patient-reported oral mucositis". | Assessed at the 8th, 15th and the 21st day after application of the interventions.
  Primary outcome is measured using Children International Mucostitis Evaluation Scale (CHIMES).ChIMES1-4 each received a score of 0-5 where 5 is the worst degree of symptoms. ChIMES5 and ChIMES6 received a score of 1 or 0 if the child had received pain medications or not. Finally, ChIMES7 received a score of 1or 0 if oral ulcers were present or not. Any question that was scored as missing or 'I can't tell' was excluded from the total possible score. If all the questions were answered, the maximum score was 23. The ChIMES Total Score was the sum of all scores; 'I can't tell' responses and missing responses both received a score of 0. The ChIMES Percentage Score was the ChIMES Total Score over the total maximum score taking into account 'I can't tell' responses (by subtracting these items from the maximum score) multiplied by 100. Higher values indicate a worse outcome.

SECONDARY OUTCOMES:
Change in "Clinical assessment of oral mucositis". | Assessed at the 8th,15th and the 21st day after application of the interventions.
  Assessed using Oral Mucositis World Health Organization Toxicity Scale.It represents grades of oral mucositis ranging from 0-4 with higher grades indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Norhan A Eldokkky, PHD, Study Director — Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided